CLINICAL TRIAL: NCT06856421
Title: Auricular Acupressure for Perimenopausal Insomnia: A Multicenter Randomized Controlled Clinical Trial
Brief Title: Auricular Acupressure for Perimenopausal Insomnia
Acronym: Acupressure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Howest (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KLS-610-01; 2024-KLS-610-01 (Registry Identifier: Ethical Review Approval)
Record Dates: First submitted 2025-02-10; First posted 2025-03-04 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Perimenopausal Insomnia
Keywords: Perimenopausal Insomnia; Auricular point

STUDY DESIGN:
Intervention Model Description: Perimenopausal insomnia patients
Who Masked: Participant, Investigator
Masking Description: To maintain blinding integrity throughout the trial duration, all participants, clinical outcome assessors, and data analysts will remain blinded to treatment allocation. In instances requiring concurrent treatment sessions, patients will undergo staggered screening processes and be assigned to separate isolated treatment rooms, thereby eliminating potential inter-participant communication that could inadvertently compromise blinding efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ear Acupoint Pressing Group (Experimental): Auricular point compression
  Interventions: Behavioral: Auricular point compression
- Sham Ear Acupoint Pressing Group (Sham Comparator): patients in this group do not perform acupoint stimulation as part of their treatment.
  Interventions: Behavioral: No pressure on the ear point

INTERVENTIONS:
Behavioral: Auricular point compression — Acupuncture Points: Endocrine, Sympathetic, Shenmen, Heart
  Procedure Instructions:
  Disinfect the areas with 75% alcohol as per standard precautions. Treatments use only ear patches without Vaccaria seeds applied to these specific acupuncture points.
  Treatment sessions occur every Monday and Thursday. On Mondays, left ears are patched for three continuous days. Then on Thursdays, qualified medical personnel will remove the patches from the left ear and apply new patches to the right ear for four consecutive days. Any replacements must be performed at the hospital by qualified staff; patients should not attempt to do this themselves.
  This procedure is repeated weekly over a span of four weeks, resulting in eight total applications. Importantly, patients in this group do not perform acupoint stimulation as part of their treatment.
  Arms: Ear Acupoint Pressing Group
Behavioral: No pressure on the ear point — Acupuncture Points: Endocrine, Sympathetic, Shenmen, Heart
  Procedure Instructions:
  Disinfect the areas with 75% alcohol as per standard precautions. Treatments use only ear patches without Vaccaria seeds applied to these specific acupuncture points.
  Treatment sessions occur every Monday and Thursday. On Mondays, left ears are patched for three continuous days. Then on Thursdays, qualified medical personnel will remove the patches from the left ear and apply new patches to the right ear for four consecutive days. Any replacements must be performed at the hospital by qualified staff; patients should not attempt to do this themselves.
  This procedure is repeated weekly over a span of four weeks, resulting in eight total applications. Importantly, patients in this group do not perform acupoint stimulation as part of their treatment.
  Arms: Sham Ear Acupoint Pressing Group

SUMMARY:
This clinical trial aims to determine whether auricular Acupressure therapy can improve symptomatic insomnia in perimenopausal women.

Can ear acupressure therapy significantly improve sleep quality in perimenopausal women with insomnia? What medical issues or adverse reactions might participants experience during the treatment? Researchers will compare ear acupressure therapy with traditional treatments in a control group to assess its effectiveness and safety.

Participants will:

Receive auricular acupressure on Monday and Thursday, applying pressure for 3 consecutive days each week. This process will continue for 4 weeks, totaling 8 sessions.

Record assessment points as follows: Baseline (2 weeks before treatment to Week 0), mid-treatment (2 weeks after treatment begins), end of treatment (4 weeks after treatment begins), and follow-up (4 weeks after treatment ends) for primary and secondary outcome indicators. Eight weeks after treatment concludes, only the primary outcome indicator (Insomnia Severity Index) will be recorded.

This trial seeks to evaluate the potential benefits and safety profile of auricular acupressure therapy for managing insomnia in perimenopausal women.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled clinical trial. Perimenopausal insomnia patients will be randomly assigned to the ear acupoint pressing group or the sham ear acupoint pressing group in a 1:1 ratio.

2.2 Randomization and Blinding Sequence Generation

* Allocation ratio: 1:1 randomization between groups
* Randomized groups: Genuine auricular acupressure group vs. Sham auricular acupressure group
* Randomization tool: SAS software version 9.3 (SAS Institute Inc.)
* Sequence generation: Performed by an independent statistician with no involvement in trial execution or statistical analysis Allocation Concealment Mechanism
* Sequence storage: Secured in a dedicated randomization sequence management system inaccessible to study personnel
* Implementation: Centralized web-based randomization system assigns participants with equal probability after baseline assessments
* Coordination: Clinical research coordinators initiate randomization requests Blinding Procedures
* Blinded parties: Participants, outcome assessors, and statisticians remain blinded to group assignments
* Treatment isolation: Concurrent treatments for ≥2 participants conducted in separate rooms to prevent cross-communication
* Data confidentiality: Intervention details withheld until final statistical analysis completion
* Blind maintenance: Comprehensive measures implemented to preserve blinding integrity
* Emergency unblinding:

Permitted only for acute medical emergencies requiring urgent clinical management Unblinded participants discontinued from efficacy analysis but retained in safety datasets Alternative therapeutic options provided to affected participants • Ethical disclosure: Participants informed about two distinct intervention arms while maintaining blinding integrity

Training:

Acupuncture doctors supervising medical staff at various centers will provide training on techniques, ensuring uniform implementation across all sites.

2.3 Blinding Assessment for Assessors and Participants Data Collection

* Administer post-treatment questionnaires to participants and assessors to document perceived group assignments Blinding Indices Calculation
* James Blinding Index (JBI):

Range: 0 (complete unblinding) to 1 (perfect blinding) Blinding failure threshold: Two-sided confidence interval upper limit <0.5

• Bang Blinding Index (BBI): Range: -1 (ideal blinding) to 1 (complete unblinding) Blinding failure threshold: One-sided confidence interval excludes 0 Statistical Implementation

* Analysis performed using R statistical software (version ≥4.2.0) for index calculations and confidence interval estimation Interpretation & Reporting
* Investigate root causes if indices suggest compromised blinding
* Full documentation of methodology, results, and conclusions in clinical study reports Emergency Unblinding Protocol
* Strict adherence to predefined Standard Operating Procedures (SOPs) for urgent unmasking scenarios Blinding Quality Assurance
* Regular monitoring/auditing of blinding integrity
* Preventive measures against accidental unmasking

Evaluation Indicators:

Primary Outcome: Insomnia Severity Index (ISI) Secondary Outcomes: Pittsburgh Sleep Quality Index (PSQI), Sleep Diary, Kupperman Index (KI), Menopause-Specific Quality of Life (MENQOL), Heart Rate Variability (HRV)

Emergency Medication:

Eszopiclone (Pharmaceutical Co., Ltd, China) will be used as emergency medication under the guidance of a psychiatric expert. The usage frequency, dosage, number of patients, and administration details during the trial will be recorded for subsequent analysis.

Follow-Up: Follow-up assessments will take place at 4 weeks post-treatment for secondary outcomes and at 8 weeks post-treatment for ISI (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 55 years;

  * Meetingperimenopause defined by the Staging of Reproductive Aging Workshop (STRAW);

    * Patients must satisfy at least one diagnostic criterion for insomnia in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5); ④ Nighttime sleep disturbances and associated perimenopausal symptoms persisting for at least 4 weeks; ⑤ No use, or stable long-term use (>2 months) of medications for treating insomnia;

      * No prior auricular acupuncture therapy, good compliance, understanding of the study protocol, and signed informed consent.

Exclusion Criteria:

* Does not meet inclusion criteria;

  * Non-natural menopausal transition due to premature ovarian failure, drug intake, or surgeries (e.g., oophorectomy);

    * Currently pregnant or breastfeeding;

      * Insomnia caused by systemic diseases (e.g., stroke, Parkinson's disease, surgery, etc.);

        * Presence of insomnia symptoms before the perimenopausal period;

          * Infection in the areas near selected acupoints; ⑦ History of alcohol or substance abuse/addiction；

            * Co-existing mental or psychological disorders (e.g., depression, generalized anxiety disorder, bipolar disorder, obsessive-compulsive disorder, etc.) or suicidal tendencies, in addition to insomnia; ⑨ Receipt of auricular acupuncture therapy within the past 3 months; ⑩ Participation in other clinical trials in the past 3 months;

              * Any known chronic pain disorders that could affect sleep.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severe Index | Baseline (2 weeks before treatment), pre-treatment (0 days of treatment), mid-treatment (2 weeks after start of treatment), end of treatment (4 weeks after start of treatment), follow-up (4 weeks and 8 weeks after end of treatment）、
  The ISI (Insomnia Severity Index) is a widely used self-assessment tool for evaluating the severity of insomnia. Its total score categorizes the severity of insomnia into four levels: no significant clinical insomnia (0-7 points), mild insomnia (8-14 points), moderate clinical insomnia (15-21 points), and severe clinical insomnia (22-28 points). The internal consistency of the ISI is Cronbach's α = 0.76, indicating good reliability. It is highly sensitive to changes after auricular acupuncture therapy, and a decrease in the ISI score of less than 8 points indicates improvement in insomnia symptoms.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | Baseline (2 weeks before treatment), pre-treatment (0 days of treatment), mid-treatment (2 weeks after start of treatment), end of treatment (4 weeks after start of treatment), follow-up (4 weeks after end of treatment
  The questionnaire examines in detail the seven key dimensions related to sleep over the past month: sleep duration, sleep disorders, latency to fall asleep, the effects of nighttime sleep on daytime function, sleep efficiency, the use of drugs needed to promote sleep, and overall sleep quality.
Sleep Diary | Baseline (2 weeks before treatment), pre-treatment (0 days of treatment), mid-treatment (2 weeks after start of treatment), end of treatment (4 weeks after start of treatment), follow-up (4 weeks after end of treatment）
  Multiple sleep parameters recorded in the sleep diary, including sleep latency, sleep efficiency, total sleep duration, and the number and duration of arousal during sleep. To comprehensively capture the participants' sleep patterns and quality changes, we asked them to fill in the sleep diary carefully daily during the 4-week intervention period and one week before each follow-up visit.
Kupperman Index | Baseline (2 weeks before treatment), pre-treatment (0 days of treatment), mid-treatment (2 weeks after start of treatment), end of treatment (4 weeks after start of treatment), follow-up (4 weeks after end of treatment）
  The KI score is currently widely used internationally to evaluate the severity of symptoms in the menopausal syndrome.
Menopause-specificquality of life | Baseline (2 weeks before treatment), pre-treatment (0 days of treatment), mid-treatment (2 weeks after start of treatment), end of treatment (4 weeks after start of treatment), follow-up (4 weeks and 8 weeks after end of treatment）、
  MENQOL Scale (total score of 174 points), different from the Kupperman score, patients should fill it out by themselves, and monitor the severity and progression of their symptoms in real time based on their own feelings.
Heart Rate Variability | Baseline (2 weeks before treatment), pre-treatment (0 days of treatment), mid-treatment (2 weeks after start of treatment), end of treatment (4 weeks after start of treatment), follow-up (4 weeks and 8 weeks after end of treatment）、
  Also known as heart rate volatility, refers to the change of the difference of heartbeat cycle by time. By testing various indicators of individual heart rate variability, it can provide information about autonomic nervous system, pressure state and other aspects, and provide clues and basis for guiding clinical and scientific research.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2025-3-1